CLINICAL TRIAL: NCT01319045
Title: Iloprost for the Treatment of Pulmonary Hypertension in Adults With Congenital Heart Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment was too slow
Sponsor: University of California, Los Angeles (Other)
Collaborators: Actelion (Industry)
Responsible Party: Principal Investigator, Jamil Aboulhosn, Assistant Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Iloprost ACHD
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Pulmonary Arterial Hypertension; Congenital Heart Disease; Eisenmenger's Syndrome
Keywords: Pulmonary Arterial Hypertension; Congenital Heart Disease; Eisenmenger's Syndrome; Prostacyclin; Iloprost
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Defects, Congenital; Eisenmenger Complex | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iloprost (Experimental): Participants will be administered iloprost at 5 mcg/dose x 6 doses daily for 3 months.
  Interventions: Drug: Iloprost

INTERVENTIONS:
Drug: Iloprost — Aerosolized iloprost, 5 mcg/dose x 6 doses daily for 3 months
  Other Names: Ventavis, prostacyclin analogue

SUMMARY:
Pulmonary arterial hypertension (PAH), or high blood pressure in the lungs, is common in patients with congenital heart disease. Historically these patients suffered significant morbidity and mortality due to a lack of effective therapies. More recently, advanced therapies which target the mechanisms underlying the development and progression of PAH have been introduced into clinical care. Oral, intravenous, subcutaneous, and inhaled therapies are all available for the treatment of PAH. Patients with PAH are first treated with oral agents (including sildenafil and bosentan). However, if these agents fail to achieve the desired effect for the patient, intravenous or inhaled therapies may be initiated. Combination therapy with multiple agents is common in routine clinical care. However, the most efficacious therapeutic regimen has yet to be delineated. The present study seeks to evaluate the efficacy of one specific regimen: iloprost, an inhaled prostacyclin derivative, used in combination with oral therapy (sildenafil and/or bosentan). Iloprost has been approved by the FDA for use in this patient population. Adults with PAH already receiving oral therapy will be invited to participate in this study. Iloprost will be added to their current therapeutic regimen for a period of three months, with pre- and post-treatment assessments. These will include a cardiopulmonary exercise test, BNP (a blood test), six minute walking distance, and a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Congenital heart disease with pulmonary arterial hypertension and cyanosis (resting oxygen saturation < 90% on room air)
* Stable on oral therapy (PDE5 inhibitor and/or endothelin blockade) for at least three months

Exclusion Criteria:

* Age < 18 years old
* Current intravenous or subcutaneous prostacyclin therapy
* Resting Systemic Hypotension (Systolic blood pressure < 85 mmHg)
* Women who are pregnant or may become pregnant (unwilling to utilize effective contraception), as well as nursing mothers
* Inability to ambulate
* Planned surgical procedure during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamil A Aboulhosn, MD, Principal Investigator — Ahmanson / UCLA Adult Congenital Heart Disease Center
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Beghetti M, Tissot C. Pulmonary arterial hypertension in congenital heart diseases. Semin Respir Crit Care Med. 2009 Aug;30(4):421-8. doi: 10.1055/s-0029-1233311. Epub 2009 Jul 24. PMID 19634081
- [Background] Humbert M, Morrell NW, Archer SL, Stenmark KR, MacLean MR, Lang IM, Christman BW, Weir EK, Eickelberg O, Voelkel NF, Rabinovitch M. Cellular and molecular pathobiology of pulmonary arterial hypertension. J Am Coll Cardiol. 2004 Jun 16;43(12 Suppl S):13S-24S. doi: 10.1016/j.jacc.2004.02.029. PMID 15194174
- [Background] Niwa K, Perloff JK, Kaplan S, Child JS, Miner PD. Eisenmenger syndrome in adults: ventricular septal defect, truncus arteriosus, univentricular heart. J Am Coll Cardiol. 1999 Jul;34(1):223-32. doi: 10.1016/s0735-1097(99)00153-9. PMID 10400015
- [Background] Daliento L, Somerville J, Presbitero P, Menti L, Brach-Prever S, Rizzoli G, Stone S. Eisenmenger syndrome. Factors relating to deterioration and death. Eur Heart J. 1998 Dec;19(12):1845-55. doi: 10.1053/euhj.1998.1046. PMID 9886728
- [Background] Christman BW. Lipid mediator dysregulation in primary pulmonary hypertension. Chest. 1998 Sep;114(3 Suppl):205S-207S. doi: 10.1378/chest.114.3_supplement.205s. PMID 9741570
- [Background] Barst RJ, Rubin LJ, Long WA, McGoon MD, Rich S, Badesch DB, Groves BM, Tapson VF, Bourge RC, Brundage BH, Koerner SK, Langleben D, Keller CA, Murali S, Uretsky BF, Clayton LM, Jobsis MM, Blackburn SD, Shortino D, Crow JW; Primary Pulmonary Hypertension Study Group. A comparison of continuous intravenous epoprostenol (prostacyclin) with conventional therapy for primary pulmonary hypertension. N Engl J Med. 1996 Feb 1;334(5):296-301. doi: 10.1056/NEJM199602013340504. PMID 8532025
- [Background] Badesch DB, Tapson VF, McGoon MD, Brundage BH, Rubin LJ, Wigley FM, Rich S, Barst RJ, Barrett PS, Kral KM, Jobsis MM, Loyd JE, Murali S, Frost A, Girgis R, Bourge RC, Ralph DD, Elliott CG, Hill NS, Langleben D, Schilz RJ, McLaughlin VV, Robbins IM, Groves BM, Shapiro S, Medsger TA Jr. Continuous intravenous epoprostenol for pulmonary hypertension due to the scleroderma spectrum of disease. A randomized, controlled trial. Ann Intern Med. 2000 Mar 21;132(6):425-34. doi: 10.7326/0003-4819-132-6-200003210-00002. PMID 10733441
- [Background] Simonneau G, Barst RJ, Galie N, Naeije R, Rich S, Bourge RC, Keogh A, Oudiz R, Frost A, Blackburn SD, Crow JW, Rubin LJ; Treprostinil Study Group. Continuous subcutaneous infusion of treprostinil, a prostacyclin analogue, in patients with pulmonary arterial hypertension: a double-blind, randomized, placebo-controlled trial. Am J Respir Crit Care Med. 2002 Mar 15;165(6):800-4. doi: 10.1164/ajrccm.165.6.2106079. PMID 11897647
- [Background] Olschewski H, Simonneau G, Galie N, Higenbottam T, Naeije R, Rubin LJ, Nikkho S, Speich R, Hoeper MM, Behr J, Winkler J, Sitbon O, Popov W, Ghofrani HA, Manes A, Kiely DG, Ewert R, Meyer A, Corris PA, Delcroix M, Gomez-Sanchez M, Siedentop H, Seeger W; Aerosolized Iloprost Randomized Study Group. Inhaled iloprost for severe pulmonary hypertension. N Engl J Med. 2002 Aug 1;347(5):322-9. doi: 10.1056/NEJMoa020204. PMID 12151469
- [Background] McLaughlin VV, Oudiz RJ, Frost A, Tapson VF, Murali S, Channick RN, Badesch DB, Barst RJ, Hsu HH, Rubin LJ. Randomized study of adding inhaled iloprost to existing bosentan in pulmonary arterial hypertension. Am J Respir Crit Care Med. 2006 Dec 1;174(11):1257-63. doi: 10.1164/rccm.200603-358OC. Epub 2006 Aug 31. PMID 16946127
- [Background] Krug S, Sablotzki A, Hammerschmidt S, Wirtz H, Seyfarth HJ. Inhaled iloprost for the control of pulmonary hypertension. Vasc Health Risk Manag. 2009;5(1):465-74. doi: 10.2147/vhrm.s3223. PMID 19475782
- [Background] Hallioglu O, Dilber E, Celiker A. Comparison of acute hemodynamic effects of aerosolized and intravenous iloprost in secondary pulmonary hypertension in children with congenital heart disease. Am J Cardiol. 2003 Oct 15;92(8):1007-9. doi: 10.1016/s0002-9149(03)00991-3. PMID 14556887
- [Background] Limsuwan A, Khosithseth A, Wanichkul S, Khowsathit P. Aerosolized iloprost for pulmonary vasoreactivity testing in children with long-standing pulmonary hypertension related to congenital heart disease. Catheter Cardiovasc Interv. 2009 Jan 1;73(1):98-104. doi: 10.1002/ccd.21793. PMID 19089967

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iloprost
Started | 5
Completed | 3 (Study was discontinued due to low enrollment)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Iloprost
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of Participants with adverse events, specifically mortality and heart failure.
Time Frame: 3 months
Population: Number of adverse events.
Measure: Number; unit: participants
Arm/Group | Iloprost
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: Exercise Capacity
Description: Change in exercise duration (modified Bruce protocol), maximal oxygen consumption (VO2 max), and/or VE/VCO2 ratio.
Time Frame: 3 months
Population: unable to analyze because study was terminated prematurely and therefore follow up assessments were not obtained
Arm/Group | Iloprost
Number analyzed (Participants) | 0

3. Secondary Outcome: Serum Brain Natriuretic Peptide (BNP)
Description: Change in serum BNP level
Time Frame: 3 months
Population: unable to analyze because study was terminated prematurely and therefore follow up assessments were not obtained
Arm/Group | Iloprost
Number analyzed (Participants) | 0

4. Secondary Outcome: Quality of Life
Description: Change in quality of life as assessed by SF-36 QOL
Time Frame: 3 months
Population: unable to analyze because study was terminated prematurely and therefore follow up assessments were not obtained
Arm/Group | Iloprost
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Iloprost
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Enrollment was too slow. The trial was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No